CLINICAL TRIAL: NCT07009431
Title: MHLDA Nursing Associates Focus Group
Status: Completed | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2425.RCHT.50
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Focus Group Study of UK Nursing and Midwifery Council Registrant Nursing Associates Working in Mental Health, Learning Disability and Autism Services
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Focus group study of UK Nursing and Midwifery Council registrant nursing associates working in mental health, learning disability and autism services

DETAILED DESCRIPTION:
This qualitative, contextual study seeks to subject data generated from focus groups to thematic analysis. A survey population of Nursing and Midwifery Council registrant nursing associates working in mental health, learning disability and autism services will be recruited via social media and professional networks. Ethical protocols will be observed during the recruitment process and beyond. Focus group cohort members will be allocated to a specific focus group session. Focus group participation will be limited to one session per volunteer. Participants will be invited to discuss their views, ideas and responses to various questions designed to reflect the research questions and objectives. Focus groups will be conducted via Microsoft Teams. Focus group discussions will be recorded and transcribed, the transcripts will be subjected to thematic analysis. Thematic analysis of focus group transcripts will be conducted using NVivo software (version 15), licensed to the Chief Investigators and Study Sponsors employing organisation (Royal Cornwall Hospitals Trust). Post focus group a follow up email will will be sent to all participants containing a summary of the topics of discussion, confirmation that their focus group participation has been completed and the proposed schedule for publishing the final report, of which they will sent a copy.

ELIGIBILITY:
Inclusion Criteria:

* Registered Nursing Associates (Nursing and Midwifery Council).
* Employed in NHS; mental health, learning disability or autism services in England.

Exclusion Criteria:

* Non-registered nursing associates.
* Trainee or student nursing associates.
* Registered nursing associates practicing in non MHLDA service.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Registered Nursing Associates (Nursing and Midwifery Council).employed in NHS; mental health, learning disability or autism services in England.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
To present a descriptive representation of the MHLDA nursing associates experience within the context of professional identity and themes reflective of nursing in their care setting | 3 months
  To understand the experiences of NAs working in MHLDA settings in the NHS through focus group sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Cornwall Hospitals Trust, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No